CLINICAL TRIAL: NCT06184711
Title: Efficiency of McNeill Dysphagia Therapy Program Combined With Transcranial Magnetic Stimulation in Individuals With Post-Stroke Dysphagia
Brief Title: McNeill Dysphagia Therapy Program Combined With Transcranial Magnetic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Kübra Nur Şimşek, Speech and Language Therapist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraCHBilkentKNS
Record Dates: First submitted 2023-12-11; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial Magnetic Stimulation combined with the McNeill Dysphagia Therapy Programme (Experimental): The McNeill Dysphagia Therapy programme (MDTP) combined with Transcranial Magnetic Stimulation (TMS) will be applied to the first experimental group.
  Interventions: Device: Transcranial Magnetic Stimulation+McNeill Dysphagia Therapy Programme
- Sham Transcranial Magnetic Stimulation combined with the McNeill Dysphagia Therapy programme (Sham Comparator): The McNeill Dysphagia Therapy programme (MDTP) combined with sham Transcranial Magnetic Stimulation (TMS) will be applied to the sham comparator group.
  Interventions: Device: Sham Transcranial Magnetic Stimulation +McNeill Dysphagia Therapy Programme
- Transcranial Magnetic Stimülation (Experimental): Only Transcranial Magnetic Stimulation (TMS) will be applied to the second experimental group.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation+McNeill Dysphagia Therapy Programme — The McNeill Dysphagia Therapy programme (MDTP) combined with Transcranial Magnetic Stimulation (TMS) will be applied to the first experimental group.
  Arms: Transcranial Magnetic Stimulation combined with the McNeill Dysphagia Therapy Programme
Device: Sham Transcranial Magnetic Stimulation +McNeill Dysphagia Therapy Programme — The McNeill Dysphagia Therapy programme (MDTP) combined with sham Transcranial Magnetic Stimulation (TMS) will be applied to the sham comparator group.
  Arms: Sham Transcranial Magnetic Stimulation combined with the McNeill Dysphagia Therapy programme
Device: Transcranial Magnetic Stimulation — Only Transcranial Magnetic Stimulation (TMS) will be applied to the second experimental group.
  Arms: Transcranial Magnetic Stimülation

SUMMARY:
This study aimed to investigate the effectiveness of the McNeill Dysphagia Therapy (MDTP) programme combined with Transcranial Magnetic Stimulation (TMS) in individuals with post-stroke dysphagia.

DETAILED DESCRIPTION:
Stroke is a neurological disorder that causes focal or global cerebral dysfunction caused by vascular causes, can last for 24 hours or longer, or may result in death. Many complications occur after stroke, and one of the most common complications is dysphagia After dysphagia, individuals with dehydration, malnutrition, aspiration, aspiration-related pneumonia, sepsis, and even death may result if no precautions are taken. Purpose of dysphagia treatment; It is to ensure that individuals receive their daily water and calorie needs most reliably. Another goal is to switch the patient to oral nutrition as much as possible. McNeill Dysphagia Therapy Programme is a systematic exercise-based therapy program developed for individuals with dysphagia. It is also frequently used in the rehabilitation of stroke, traumatic brain injury, and post-cancer dysphagia. Transcranial Magnetic Stimulation (TMS) is based on the principle of electromagnetic induction. It is a non-invasive method that, together with the magnetic field created by a coil placed on the scalp, causes electrical stimulation in the cerebral cortex and creates neurophysiological arrangements in different parts of the brain. Without the electrode, electrical energy is transferred to the human brain and the cerebral cortex is stimulated. An action potential is created by stimulation in neuronal membranes and causes neurons to fire. Thus, nerve cells are stimulated and the process of reorganization of the brain begins. With the stimulation of the cerebral cortex, the swallowing centre is stimulated and the muscles associated with swallowing are activated. The efficacy of MDTP combined with r TMS, MDTP combined with sham r TMS and r TMS alone will be compared in the intervention of dysphagia after stroke. Patients in all three groups will be subjected to both clinical assessment tools and instrumental evaluation before and after treatment. Data will be evaluated using the Mann Swallowing Ability Assessment Test, Penetration Aspiration Scale, Functional Oral Intake Scale, Visual Analogue Scale, Dynamic Rating Scale of Swallowing Toxicity, Dysphagia Severity Rating Scale

ELIGIBILITY:
Inclusion Criteria:

Dysphagia Diagnosis of ischaemic stroke Over 18 years old Cognitively competent and co-operative

Exclusion Criteria:

Epilepsy or seizure risk record Carry metallic objects in the head (such as arterial clips, plates, screws), eye or brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-29 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Change from baseline from 3 weeks
  Penetration Aspiration Scale (PAS): An 8-point severity rating. Scale 1 = no substance enters the airways 8 = substance enters the airways, passes under the vocal cords without any effort to expel it.
Functional Oral Intake Scale | Change from baseline from 3 weeks
  FOIS is a scale ranging from 1 (nothing by mouth) to 7 (total oral diet with no restriction)
Dynamic Rating Scale of Swallowing Toxicity | Change from baseline from 3 weeks
  Dynamic Imaging Grading of Ingestion Toxicity (DIGEST): residue less than 10% of the bolus = 0 point, residue less than half of the bolus = 1 point, residue less than 90% of the bolus = 2 points, residue more than 90% of the bolus = 3 points, residue in all consistencies tested = 4 points.
Dysphagia Severity Scale | Change from baseline from 3 weeks
  Dysphagia Severity Scale (DSS); those ranked from "level 1" to "level 4'' are categorized into the "choking/aspiration group (severe group)". In DSS, those ranked from "level 5" to "level 7'' are categorized into the "without choking/aspiration group (mild group)".

SECONDARY OUTCOMES:
Mann Swallowing Ability Assessment Test | Change from baseline from 3 weeks
  It is used for the assessment of oro-motor/sensory prerequisite skills of swallowing, functional assessment of swallowing and dietary modifications and identification of risk factors. A score of 138 and below indicates severe dysphagia, 139-167 indicates moderate dysphagia, 168-177 indicates mild dysphagia and 178-200 indicates no abnormality in swallowing.
Visual Analogue Scale (VAS) | Change from baseline from 3 weeks
  Visual Analogue Scale; Line bisection task or numerical grading.The patient 'marks' the point of current swallowing ability. He/she scores his/her swallowing from 1 to 10.
  - The patient 'marks' the point of current swallowing ability. He/she scores his/her swallowing from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Nur ŞİMŞEK, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)